CLINICAL TRIAL: NCT06700577
Title: Prevalence of Multidrug Resistant Tuberculosis by Xpert MTB/RIF Ultra and Xpert XDR Assay Among Newly Diagnosed Cases
Brief Title: Multidrug Resistance in Newly Diagnosed TB Patient
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma nashat esmail zyada, Pulomongist , principale investigator , Resident doctor, Assiut University
Other Study IDs: Gene expert and Tuberculosis
Record Dates: First submitted 2024-09-14; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Gene expert — Gene expert and XDR to detect multidrug resistance between tb patient
Genetic: Ultra xpert and xdr xpert — Detect resistance between tyberculous patient

SUMMARY:
Tuberculosis (TB) is one of the major public health threats, competing with the human immunodeficiency virus (HIV) as the cause of death due to infectious diseases worldwide.

Multi drug-resistant Mycobacterium tuberculosis (MDR-TB) is one of the leading causes of death in the world.

The resource constraints make it difficult to diagnose and monitor the cases of MDR-TB.

GeneXpert is a recognized tool used to diagnose the patients of pulmonary tuberculosis in clinical settings across the globe MDR Multidrug-resistant tuberculosis (MDR-TB), caused by Mycobacterium tuberculosis that is resistant to both isoniazid and rifampicin with or without resistance to other drugs According to current World Health Organization and the International Union Against Tuberculosis and Lung Disease estimates, the median prevalence of MDR-TB has been 1.1% in newly diagnosed patients. The proportion, however, is considerably higher (median prevalence, 7%) in patients who have previously received anti-TB treatment.

XDR tuberculosis is caused by a strain of Mycobacterium tuberculosis resistant to isoniazid and rifampin (which defines MDR tuberculosis) in addition to any fluoroquinolone and at least one of the three following injectable drugs: capreomycin, kanamycin, and amikacin The main causes of the spread of resistant TB are weak medical Systems, amplification of resistance patterns through incorrect treatment, and transmission in communities and facilities. Although patients harboring MDR and XDR strains present a formidable challenge for treatment, cure is often possible with early identification of resistance and use of a properly designed regimen.

DETAILED DESCRIPTION:
To detect the prevalence of MDR T.B. using xpert MTB/RIF ultra and XDR assay in newly diagnosed cases

ELIGIBILITY:
Inclusion criteria

* newly diagnosed tuberculosis patient
* Diagnosed by direct smear for sputum or body fluid

Exclusion Criteria:

* previously treated patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All newly diagnosed TB patient above 18 years who not recieved antituberculus drug before
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
To detect the prevalence of multidrug resistant tuberculosis in newly diagnosed cases by xpert XDR assay. | Baseline

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Seung KJ, Keshavjee S, Rich ML. Multidrug-Resistant Tuberculosis and Extensively Drug-Resistant Tuberculosis. Cold Spring Harb Perspect Med. 2015 Apr 27;5(9):a017863. doi: 10.1101/cshperspect.a017863. PMID 25918181